CLINICAL TRIAL: NCT00090844
Title: Preservation of Ovarian Function in Young Women Treated With (Neo) Adjuvant Chemotherapy for Breast Cancer: A Randomized Trial Using the Gonadotropin-releasing Hormone (GnRH) Agonist (Triptorelin) During Chemotherapy
Brief Title: Triptorelin for Preserving Ovarian Function in Premenopausal Women Receiving Chemotherapy for Early-Stage Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early closure due to low accrual
Sponsor: University of South Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000374991; P30CA076292 (NIH); MCC-0203 (Other: Moffitt CCOP Research Base); NCI-7031 (Other: National Cancer Institute Division of Cancer Prevention)
Record Dates: First submitted 2004-09-07; First posted 2004-09-08 (Estimated); Results first posted 2013-01-21 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2013-01

CONDITIONS: Breast Cancer; Hormone Changes; Drug Toxicity
Keywords: drug/agent toxicity by tissue/organ; hormone changes; stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms; Drug-Related Side Effects and Adverse Reactions | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- triptorelin (Experimental): GnRH analogue (triptorelin) during chemotherapy
  Interventions: Drug: triptorelin
- no triptorelin (No Intervention): No GnRH analogue (triptorelin) during chemotherapy

INTERVENTIONS:
Drug: triptorelin — 3.75 mg TRELSTAR DEPOT (triptorelin) administered monthly as single intramuscular injection
  Other Names: Trelstar Depot
  Arms: triptorelin

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Chemoprotective drugs, such as triptorelin, may protect normal ovarian cells from the side effects of chemotherapy.

PURPOSE: This randomized phase II trial is studying how well triptorelin works in preserving ovarian function in premenopausal women who are receiving chemotherapy for early-stage breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the protective effect of chemical ovarian suppression using triptorelin on the preservation of ovarian function in premenopausal women with early-stage operable breast cancer undergoing adjuvant or neoadjuvant systemic chemotherapy.

Secondary

* Determine the rate of chemotherapy-related amenorrhea in patients treated with this drug.
* Determine the value of inhibin A and B as alternative markers of premature ovarian failure in patients treated with this drug.
* Determine quality of life of patients treated with this drug.
* Determine disease-free and overall survival of patients treated with this drug.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (< 35 years vs 35 to 39 years vs > 39 years); concurrent neoadjuvant or adjuvant systemic chemotherapy (fluorouracil, epirubicin, and cyclophosphamide [6 courses] OR fluorouracil, doxorubicin, and cyclophosphamide [6 courses] vs doxorubicin and cyclophosphamide [AC] [4 courses] vs doxorubicin and cyclophosphamide [AC] [4 courses] followed by a taxane [4 courses]); and hormone receptor status (estrogen receptor [ER]- AND progesterone receptor [PR]-negative vs ER- OR PR-positive).

* Arm I: Beginning within 1-4 weeks before the start of chemotherapy, patients receive triptorelin intramuscularly once monthly for 4-6 months during neoadjuvant or adjuvant systemic chemotherapy.
* Arm II: Patients receive neoadjuvant or adjuvant systemic chemotherapy only. Quality of life is assessed at baseline, monthly during treatment, every 6 months for 2 years, and then annually for 3 years.

Patients are followed every 6 months for 2 years and then annually for 3 years.

PROJECTED ACCRUAL: A total of 138 patients (69 per treatment arm) will be accrued for this study within 35 months.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer

  * Early-stage, operable disease
* Scheduled to receive adjuvant or neoadjuvant systemic chemotherapy for breast cancer
* Hormone receptor status:

  * Meets 1 of the following criteria:

    * Estrogen receptor (ER)- OR progesterone receptor (PR)-positive
    * ER- AND PR-negative
* No history of premature ovarian failure

PATIENT CHARACTERISTICS:

Age

* Under 45

Sex

* Female

Menopausal status

* Premenopausal

  * Follicle-stimulating hormone levels < 40 IU/L at baseline AND at least 2 menstrual periods within the past 6 months
* No first-degree relative menopausal at < 40 years of age

Performance status

* Eastern Cooperative Oncology Group [ECOG] 0-1

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Fertile patients must use effective non-hormonal methods of contraception
* No prior osteoporosis or other non-malignant systemic disease that would preclude prolonged follow-up
* No known allergies to gonadotrophin-releasing hormone agonists
* No other cancer except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No prior chemotherapy

Endocrine therapy

* At least 2 weeks since prior oral contraceptives
* No prior fertility treatment

  * Clomiphene or pergonal for polycystic ovarian disease allowed
* No other concurrent oral or transdermal hormonal therapy, including any of the following:

  * Estrogen
  * Progesterone
  * Androgens
  * Aromatase inhibitors
  * Hormone replacement therapy
  * Oral contraceptives

Radiotherapy

* No prior ovarian radiotherapy

Surgery

* No prior bilateral oophorectomy
* No plans for oophorectomy or hysterectomy within the next 2 years

Other

* At least 1 week since prior warfarin

Exclusion Criteria:

* History of premature ovarian failure
* Over 45 years of age
* First-degree relative menopausal at < 40 years of age
* Pregnant or nursing
* Prior osteoporosis or other non-malignant systemic disease that would preclude prolonged follow-up
* Known allergies to gonadotrophin-releasing hormone agonists
* Other cancer besides nonmelanoma skin cancer
* Prior chemotherapy
* Prior ovarian radiotherapy
* Prior bilateral oophorectomy

Max Age: 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2004-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela N. Munster, MD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (9):
- United States (9):
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - MBCCOP - JHS Hospital of Cook County, Chicago, Illinois
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - CCOP - Scott and White Hospital, Temple, Texas
  - CCOP - Northwest, Tacoma, Washington

REFERENCES:
- See also: Published Results — https://pubmed.ncbi.nlm.nih.gov/22231041/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 49 female patients were enrolled between July 2003 and January 2007.
Groups:
- Triptorelin: Gonadotropin-releasing hormone [GnRH] analogue (triptorelin) during chemotherapy
  triptorelin : 3.75 mg TRELSTAR DEPOT (triptorelin) administered monthly as single intramuscular injection
- no Triptorelin: No Gonadotropin-releasing hormone [GnRH] analogue (triptorelin) during chemotherapy
Period: Overall Study
Arm/Group | Triptorelin | no Triptorelin
Started | 27 | 22
Completed | 26 | 21
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Triptorelin | no Triptorelin | Total
Number analyzed (Participants) | 27 | 22 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 22 | 49
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 39 [21 to 44] | 38 [26 to 44] | 39 [21 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 22 | 49
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 24 | 20 | 44
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 25 | 19 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 22 | 49

OUTCOME MEASURES:

1. Primary Outcome: Time to Resumption of Menses
Description: Ovarian function as assessed by follicle stimulating hormone (FSH) and record of menses every 6 months beginning in month 6 for 2 years and then annually for 3 years
Time Frame: Baseline, end of chemotherapy then 5 years
Measure: Median (Full Range); unit: months
Groups:
- Triptorelin: GnRH analogue (triptorelin) during chemotherapy
  triptorelin : 3.75 mg TRELSTAR DEPOT (triptorelin) administered monthly as single intramuscular injection
Arm/Group | Triptorelin | no Triptorelin
Number analyzed (Participants) | 26 | 21
months | 4.96 [.43 to 28] | 5.82 [1.15 to 19]

2. Secondary Outcome: Chemotherapy-related Amenorrhea
Description: Chemotherapy-related amenorrhea as assessed by record of menses monthly during treatment. Record of menses is completed by patient throughout their time on study through chemotherapy and for 5 years.
Time Frame: Baseline, end of chemotherapy then 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Triptorelin | no Triptorelin
Number analyzed (Participants) | 26 | 21
Participants | 3 | 2

ADVERSE EVENTS:
Arm/Group | Triptorelin | no Triptorelin
Serious Adverse Events (participants affected / at risk) | 2/27 | 0/22
Other Adverse Events (participants affected / at risk) | 25/27 | 18/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triptorelin (N=27) | no Triptorelin (N=22)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0)
Febrile Neutropenia (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triptorelin (N=27) | no Triptorelin (N=22)
Fatigue (General disorders) | 4 (5) | 1 (1)
Insomnia (General disorders) | 3 (3) | 2 (2)
Sweating (diaphoresis) (General disorders) | 4 (4) | 5 (6)
Weight gain (General disorders) | 3 (3) | 1 (1)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 11 (11) | 7 (7)
hot flashes/flushes (Endocrine disorders) | 23 (38) | 12 (18)
Constipation (Gastrointestinal disorders) | 4 (5) | 2 (3)
Distension/bloating, abdominal (Gastrointestinal disorders) | 3 (3) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (2) | 3 (5)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (8) | 7 (14)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2)
Infection - Other (Infections and infestations) | 2 (2) | 2 (2)
Edema - limb (Blood and lymphatic system disorders) | 1 (1) | 2 (3)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 6 (7) | 5 (5)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 3 (4) | 3 (3)
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (4) | 0 (0)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 9 (22) | 8 (14)
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 6 (10) | 0 (0)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Mood alteration (Nervous system disorders) | 13 (15) | 6 (8)
Neuropathy: sensory (Nervous system disorders) | 2 (2) | 2 (2)
Pain (General disorders) | 10 (31) | 7 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Vaginal discharge (non-infectious) (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Headaches (General disorders) | 6 (13) | 5 (5)
Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Mucositis/stomatitis (NOS) (Gastrointestinal disorders) | 0 (0) | 2 (2)
Infection with unknown ANC (Infections and infestations) | 4 (6) | 4 (5)
Pain - Other (General disorders) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
Study closed to accrual early due to futility

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No